CLINICAL TRIAL: NCT01620333
Title: A Randomised, Open-labelled, Single-centre, Two-period Crossover Trial Characterizing the Pharmacokinetics and Pharmacodynamics of NN-X14Mix50 and NN-X14Mix70 in Healthy Male Subjects
Brief Title: Pharmacokinetics of Biphasic Insulin Aspart 50 and 70 in Japanese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1164
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment period 1 (Experimental)
  Interventions: Drug: biphasic insulin aspart 50; Drug: biphasic insulin aspart 70
- Treatment period 2 (Experimental)
  Interventions: Drug: biphasic insulin aspart 50; Drug: biphasic insulin aspart 70

INTERVENTIONS:
Drug: biphasic insulin aspart 50 — A single dose of 0.08 U/kg body weight, administered subcutaneously (s.c., under the skin) on two dosing visits in random order separated by 6-12 days
Drug: biphasic insulin aspart 70 — A single dose of 0.08 U/kg body weight, administered subcutaneously (s.c., under the skin) on two dosing visits in random order separated by 6-12 days

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to investigate the pharmacokinetics of biphasic insulin aspart 50 (NN-X14Mix50) and biphasic insulin aspart 70 (NN-X14Mix70) in Japanese healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Japanese
* Body Mass Index (BMI) of 19-27 kg/m^2 (both inclusive)
* Fasting blood glucose between 3.8-6 mmol/L (68.4-108.0 mg/dL) (both inclusive
* Considered generally healthy upon completion of medical history and physical examination, as judged by the Investigator or Sub-Investigator

Exclusion Criteria:

* Clinically significant abnormal haematology or biochemistry screening tests, as judged by the Investigator or Sub-Investigator(s)
* Any serious systemic infectious disease that occurred during the 4 weeks prior to the screening, as judged by the Investigator or Sub-Investigator
* Any inter-current illness that may affect blood glucose, as judged by the Investigator or Sub-Investigator
* Hepatitis B or C, or HIV (human immunodeficiency virus)
* Use of prescription drugs within 2 weeks preceding the screening
* Use of non-prescription drugs, except routine vitamins or drugs that may not
* Blood donation of more than 1150 mL within the last 12 months
* Subjects with a first degree relative with diabetes mellitus
* History of or presence of diabetes
* History of or presence of cancer or any clinically significant cardiac, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, dermatological, venereal, haematologic, neurologic, or psychiatric diseases or disorder
* Previous history of serious allergy or anaphylactic reaction
* Subjects who consume more than 28 units of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse
* Subjects who smoke more than 5 cigarettes per day

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2000-02; Primary Completion 2000-04 (Actual); Study Completion 2000-04 (Actual)

PRIMARY OUTCOMES:
Area under the insulin aspart curve in the interval from 0 to 24 hours (BIAsp 70)

SECONDARY OUTCOMES:
Cmax, maximum insulin aspart concentration
tmax, time to maximum insulin aspart concentration
t½, terminal elimination half life
Mean residence time (MRT)
Area under the curve from time 0 to infinity (0-∞)
Area under the insulin aspart curve in the interval from 0 to 24 hours (BIAsp 50)
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Irie S, Furuie H, Matsuguma K, Matsumura Y. Pharmacokinetics and pharmacodynamics of biphasic insulin aspart 50 and biphasic insulin aspart 70 in healthy Japanese subjects. Diabetologia 2006; 49 (Suppl 1): 612
- [Result] Irie S, Matsumura Y, Furuie H, Matsuguma K. Comparison of the pharmacokinetic and pharmacodynamic properties of biphasic insulin aspart 50 and biphasic insulin aspart 70 in healthy Japanese. Diabetic Medicine 2006; 23 (Suppl 4): 331 (P915)
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com